CLINICAL TRIAL: NCT06466369
Title: Efficacy and Safety of Once Daily Administration Tadalafil in Patients With Benign Prostatic Hyperplasia
Brief Title: Administration of Tadalafil in Patients With Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, ahmed salah saad abomandour, Principal Investigator, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 461
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: BPH With Other Lower Urinary Tract Symptoms
MeSH Terms: interventions — Tadalafil

STUDY DESIGN:
Intervention Model Description: Parallel, double-blinded, prospective, randomized controlled study.
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled group (No Intervention)
- Low-dose intervention group (Experimental)
  Interventions: Drug: Tadalafil
- High-dose intervention group (Experimental)
  Interventions: Drug: Tadalafil

INTERVENTIONS:
Drug: Tadalafil — tadalafil 2.5 mg, 5 mg
  Arms: High-dose intervention group; Low-dose intervention group

SUMMARY:
The aim of the present study is to evaluate the efficacy and safety of once daily administration PDE5 inhibitors, tadalafil for 3 months as anti-inflammatory, antiproliferative and relaxant effects in ED with BPH patients.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 45 years and sexually active with symptomatic benign prostatic hyperplasia (no hospitalization 3 months prior to start of treatment).

Exclusion Criteria:

* 1. Patients with bladder or prostate malignancy. 2. A history of lower urinary tract surgery. 3. History of catheterization. 4. Urinary retention. 5. Urinary tract infection. 6. Stone disease. 7. Any neurological disease.

Min Age: 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Evaluation of International prostate symptom score (IPSS)/quality of life (QoL). | 3 months compared to baseline
Evaluation of International index of erectile function (IIEF). | 3 months compared to baseline

CONTACTS AND LOCATIONS:
Locations (1):
- outpatient clinic of the urology department at AlZahraa University Hospital, Al-Azhar University, Faculty of Medicine for Girls., Cairo, Egypt